CLINICAL TRIAL: NCT03008603
Title: Evaluation of the Safety, Effectiveness & Usability of the XACT Robotic System for Image Guided Percutaneous Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xact Robotics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-001-00
Record Dates: First submitted 2016-12-28; First posted 2017-01-02 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: CT-guided Minimally Invasive Procedures e.g., Biopsies
Keywords: CT-guided minimally invasive procedures; Robot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Procedures with XACT Robotic System (Experimental): CT-guided minimally invasive percutaneous procedures using the XACT Robotics system
  Interventions: Device: XACT Robotic System

INTERVENTIONS:
Device: XACT Robotic System — The XACT device is a real-time, CT image guided, 3-dimensional robotic system. The XACT device is intended for use as an image guided positioning and steering system for insertion of clinical tools, such as biopsy needles, ablation needles, etc., during minimally invasive percutaneous procedures. The system is defined to guide (i.e., position and steer) the tool according to a predefined trajectory following a registration process between the device's coordinate system and real-time CT images.

SUMMARY:
This is a prospective, single-arm study is to evaluate the safety, effectiveness and usability of the XACT device. Subjects undergoing CT-guided, minimally invasive percutaneous procedures in the interventional radiology suite, e.g., core biopsy, will participate in the summary. Clinical accuracy will be the primary efficacy endpoint. Usability and safety will also be evaluated.

DETAILED DESCRIPTION:
This is a prospective, single-arm study is to evaluate the safety, effectiveness and usability of the XACT device. The study will be approved by the Institutional Review Board (IRB) at each of the participating centers prior to patient enrollment.

Subjects undergoing CT-guided, minimally invasive percutaneous procedures in the interventional radiology suite, e.g., core biopsy, fine needle aspiration (FNA), tumor ablation, etc., and willing to sign an informed consent document will be screened for compliance with the study inclusion and exclusion criteria.

A total of thirty (85) subjects will be enrolled in the study at 5 medical centers. The intention is to recruit subjects, which will cover a variety of CT-guided interventional procedures and a variety of different procedural tools that may be used with the device. Investigators will screen patients based on the inclusion/exclusion criteria described below and the subjects' demographic, general medical history, medical condition/indication, coagulation factors, concomitant medications and vital signs will be obtained.

Clinical accuracy will be the primary efficacy endpoint and is defined as the ability to place the instrument or procedural tool at a location suitable for the planned intervention. The investigator will review the final instrument position on the post-placement CT images to determine if the pre-operative planned target was reached. This information will be used to calculate success rate.

Additionally, the usability of the XACT device will be evaluated using a rating scale by assessing the ease of device setup, device operation, pre-operative planning, robot positioning, guiding and needle advancement. The total time of the procedure will be recorded, as will the number of CT scans performed and the radiation dose (DLP and CTDI). The distance from the tip of the needle/tool to the target, once the XACT robot reaches the pre-defined target will be measured in order to determine system accuracy in quantitative terms using the system tools.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Subjects undergoing CT-guided, minimally invasive percutaneous procedures in the interventional radiology suite, e.g., core biopsy, fine needle aspiration (FNA), tumor ablation, etc.
* Subject is capable and willing to provide informed consent.
* Subject is capable and willing to adhere to the study procedures

Exclusion Criteria:

* Subjects in whom the target is written 1 cm of a major blood vessel or major nerve.
* Subject with lesions in the central and peripheral nervous system and the spine.
* Subject with significant coagulopathy
* Subjects with a preexisting conditions, which, in the opinion of the investigator, may interfere with the conduct of the study
* Subjects with an unstable medical condition, e.g. unstable hypertension, unstable cardiac disease, etc.
* Subjects who are uncooperative or cannot follow instructions
* Subjects with a mental state that may preclude completion of the study procedure
* Female subjects who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is to evaluate the clinical accuracy of the XACT system. | End of procedure
  Clinical accuracy of the study will be determined by the ability of the XACT system to reach the pre-defined target in each procedure.

SECONDARY OUTCOMES:
The secondary endpoint of the study is to evaluate the usability of the XACT system under actual use clinical conditions. | End of procedure
  usability of the XACT device will be evaluated using a rating scale by assessing the ease of device setup, device operation, pre-operative planning, robot positioning, guiding and needle advancement.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | End of procedure
  Safety of the XACT device will also be evaluated by reporting the incidence, severity and frequency of all Adverse Events (AE), related and unrelated to the device treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No